CLINICAL TRIAL: NCT05807893
Title: A Multicenter, Single-arm, Open Study to Evaluate the Safety and Efficacy of Serplulimab in Combination With Bevacizumab and First-line Chemotherapy in Driver Negative Non-squamous NSCLC Patients With Brain Metastases
Brief Title: Study to Evaluate the Safety and Efficacy of Serplulimab Plus Bevacizumab and Chemotherapy in NSCLC Patients With Brain Metastases
Acronym: SUPER BRAIN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Professor of Medicine, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT27
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer Stage II; Bevacizumab; Immunotherapy; Brain Metastases
Keywords: bevacizumab; Serplulimab; efficacy; non-small cell lung cancer; brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab combined with bevacizumab and first-line chemotherapy (Experimental): Serplulimab combined with bevacizumab and first-line chemotherapy
  Interventions: Drug: Serplulimab combined with bevacizumab and first-line chemotherapy

INTERVENTIONS:
Drug: Serplulimab combined with bevacizumab and first-line chemotherapy — Serplulimab combined with bevacizumab and first-line chemotherapy

SUMMARY:
A multicenter, single-arm, open study to evaluate the safety and efficacy of Serplulimab in combination with bevacizumab and first-line chemotherapy in driver negative non-squamous NSCLC patients with brain metastases

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open study. Thirty patients with stage IV nsqNSCLC with BMs confirmed by histopathology or cytology and reported negative driver genes within three months were enrolled. To evaluate the safety, tolerability and efficacy of Serplulimab combined with bevacizumab and first-line chemotherapy in driver negative nsqNSCLC subjects with brain metastases.

Qualified subjects were selected and entered into the study in sequence. The trial was divided into combination chemotherapy period (C1-C4/C6) and maintenance treatment period (C5/C7-C32). In combination chemotherapy period, all subjects were treated with Serplulimab combined with bevacizumab and chemotherapy agents after entering the study, and in maintenance treatment period, Serplulimab combined with bevacizumab and pemetrexed. The efficacy was evaluated every 3 weeks (Q3W), every 2 cycles in combination chemotherapy and every 3 cycles in maintenance treatment. All subjects received treatment until subjects withdrew their informed consent, disease progression, intolerable toxicity, investigator judgment that medication must be discontinued, loss of follow-up, death, or 2 years of use of Serplulimab, whichever occurred first; At the end of treatment, patients were followed up for survival until death.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stage IV non-squamous non-small cell lung cancer (nsqNSCLC) with brain metastases confirmed by histopathology or cytology;
* The patient should provide a gene test report within 3 months, and the gene report showed negative driver gene, that is, no EFGR sensitive gene mutation, no ALK or ROS1 gene fusion;
* MRI confirmed brain parenchymal metastasis with ≥3 brain lesions; Or have 1-2 brain lesions but not suitable for local treatment or refuse local treatment patients. There must be at least 1 measurable lesion with a diameter ≥5mm in the brain; Patients with local meningeal metastases were allowed, but patients with extensive meningeal metastases were not included;
* For asymptomatic BMS or BMS whose intracranial hypertension symptoms were controlled after dehydration treatment, medication could be continued at the time of enrollment or during the study period to keep symptoms stable;
* There was at least one measurable target lesion as assessed by RECIST v1.1 within 4 weeks prior to initial medication;
* The patient agrees to provide the genetic test results within 3 months; if not, the patient shall provide the tumor tissue that meets the requirements for genetic test;
* ECOG PS score is 0-1; Good functioning of vital organs

Exclusion Criteria:

* A known history of severe allergy to any monoclonal antibody (NCI-CTCAE 5.0 grade greater than 3); Or known hypersensitivity to carboplatin/pemetrexed components;
* Any active infection requiring systemic anti-infective therapy occurs within 14 days prior to initial administration;
* A history of myocardial infarction and poorly controlled arrhythmias (including QTc interval ≥450 ms in men and 470 ms in women) within 6 months prior to initial administration (QTc interval calculated by Fridericia formula); Or left ventricular ejection fraction according to NYHA standard for Grade III-IV cardiac insufficiency or color Doppler ultrasound < 50%;
* The subjects had ≥ grade 2 CTCAE peripheral neuropathy;
* The subject has uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionic calcium or calcium > 12 mg/dL or corrected serum calcium > ULN);
* Subjects with prior or screening history of interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severe impairment of lung function, which the investigators judged might interfere with the detection and management of suspected drug-related pulmonary toxicity;
* Hepatitis B patients [hepatitis B surface antigen (HBsAg) positive and detection of HBV-DNA suggests viral replication]; Or hepatitis C patients [hepatitis C virus (HCV) antibody positive and HCV-RNA test indicates viral replication]; Or syphilis screening positive (specific antibody test positive, non-specific antibody test negative and combined with clinical diagnosis confirmed as non-active infection); Or a known human immunodeficiency virus (HIV) positive history or HIV screening positive;
* Subjects have known active or suspected autoimmune diseases. Subjects in stable state who did not require systemic immunosuppressive therapy were admitted;
* Other active malignancies within 5 years or at the same time. Localized tumors that have been cured for more than 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, prostate carcinoma in situ, cervical carcinoma in situ and breast carcinoma in situ, can be included in the group.
* Those who received live or attenuated vaccines within 28 days prior to the first dose or have plans to receive such vaccines during the study period; But inactivated virus vaccines for seasonal influenza are allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-14 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
iPFS | The time from receipt of study treatment to intracranial tumor PD or to death due to any cause,whichever came first, assessed up to 60 months
  The time from receipt of study treatment to intracranial tumor PD or to death due to any cause,whichever came first,

SECONDARY OUTCOMES:
PFS | The time from receipt of study treatment to PD or to death due to any cause,whichever came first, assessed up to 60 months.
  The time from receipt of study treatment to PD or to death due to any cause,,whichever came first,
OS | The time interval between enrollment and death from any cause,,whichever came first, assessed up to 60 months.
  The time interval between enrollment and death from any cause
iORR | The number and percentage of objective response (PR+CR) of intracranial tumor at each time point after treatment, through study completion, an average of 2 year.
  The number and percentage of objective response (PR+CR) of intracranial tumor at each time point after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Likun Chen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No